CLINICAL TRIAL: NCT02899247
Title: A 5-year Clinical Trial Assessing the Effects of a Surface Sealant on Composite Resin Class I Restorations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Flavia Pardo Salata Nahsan (Other)
Responsible Party: Sponsor-Investigator, Flavia Pardo Salata Nahsan, Principal Investigator, Universidade Federal de Sergipe
Organization: Universidade Federal de Sergipe (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Un. Fed. Sergipe
Record Dates: First submitted 2016-09-04; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Definitive Restorations, Longevity
Keywords: composite resin; surface sealant

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- No Surface Sealant (Experimental): Resin composite only
  Interventions: Procedure: No surface sealant
- With surface Sealant (Active Comparator): Resin composite with surface sealant application
  Interventions: Procedure: Surface sealant

INTERVENTIONS:
Procedure: Surface sealant — Device:
  * Enamel and dentin etching with 37% phosphoric acid (Scotchbond Etchant; 3M/ESPE, St. Paul, MN, USA) for 30 s and 15 s.
  * Two coats of one-bottle adhesive (Adper TM Single Bond 2, 3M/ESPE, St. Paul, MN, USA) will be applied homogeneously to the surface with a disposable micro-brush.
  * Cavities will be restored with 2 mm increments of composite resin (Z350, 3M/ESPE, St. Paul, MN, USA)
  * 7 Days after: Finishing and polishing will be performed with fine diamond and multilaminated burs, one step polishing system Pogo (Dentsply, Caulk, USA).
  * The composite surface and 1 mm external limit will be etched with a 37% acid phosphoric and after will be covered using a nanotechnology liquid polish system (Lasting Touch, Dentsply Caulk, Milford, DE, USA).
  Arms: With surface Sealant
Procedure: No surface sealant — Device:
  * Enamel and dentin etching with 37% phosphoric acid (Scotchbond Etchant; 3M/ESPE, St. Paul, MN, USA) for 30 s and 15 s.
  * Two coats of one-bottle adhesive (Adper TM Single Bond 2, 3M/ESPE, St. Paul, MN, USA) will be applied homogeneously to the surface with a disposable micro-brush.
  * Cavities will be restored with 2 mm increments of composite resin (Z350, 3M/ESPE, St. Paul, MN, USA)
  * 7 Days after: Finishing and polishing will be performed with fine diamond and multilaminated burs, one step polishing system Pogo (Dentsply, Caulk, USA).
  Arms: No Surface Sealant

SUMMARY:
This trial, based on a split mouth and double-blind design, will evaluate the effects of a surface sealant on the clinical performance of composite resin class I restorations. According to eligibility criteria, 10 pairs of upper and lower molars or premolars will be restored with Esthet X composite resin. For each pair, one surface will be sealed with Lasting Touch surface sealant. A clinical evaluation will be performed by two experienced operators using modified USPHS (United States Public Health service) after 5 years after treatment. Data will be analyzed using the McNemar test (p < 0.05).

DETAILED DESCRIPTION:
The protocol was approved by the Human Ethics Committee (protocol number 133/2010, CAAE 0124.0.224.000.-10), and all patients will sign informed consent forms and complete a registration form prior to treatment.

The eligibility criteria for participation in the study include good oral hygiene, a class I caries lesion or unsatisfactory restoration in at least two posterior teeth (molar or premolar), a buccolingual extension, and a signed consent form. The exclusion criteria includes patients with a proximal caries lesion, the presence of periodontal disease, symptomatic restored or nonrestored teeth indicating irreversible pulpal pathology, an abnormal occlusion or the absence of antagonist teeth, exposure of pulpal tissue, and extended or large cavities.

This study will include 10 patients (aged 18 to 45 years) totaling 14 pairs of class I restorations (molars and premolars). These pairs will be randomly divided into two study groups, resulting in a split-mouth design.

A hybrid resin composite, Esthet X (Dentsply, Caulk, USA) and an etch-and-rinse two-step adhesive, AdperTM Single Bond (3M, ESPE) will be used for the composite restorations. For teeth with the surface sealant, they will be covered with Lasting Touch (Dentsply, Caulk, USA).

All cavity preparations and restorations will be performed by the same experienced operator, using rubber dam isolation. Cavity designs will be prepared using a #245 carbide bur (KG Sorensen, Cotia, SP, Brazil), which will be changed every five preparations. All enamel bordered cavity margins will be verified.

The restorative procedures will be performed using rubber dam isolation. In very deep cavities, the dentin will be covered with calcium hydroxide (Dycal; Dentsply Ind. e Com. Ltda., Petrópolis, RJ, Brazil) and resin-modified glass-ionomer cement (Vitrebond, 3M ESPE, St. Paul, MN, USA). In deep cavities dentin will be covered solely with resin-modified glass-ionomer cement.

The enamel and dentin will be etched with 37% phosphoric acid (Scotchbond Etchant; 3M/ESPE, St. Paul, MN, USA) for 30 s and 15 s, respectively. Then will be rinsed with water spray for 30 s and gently and thoroughly dried with absorbent paper for 10 s.

Two coats of one-bottle adhesive (Adper TM Single Bond 2, 3M/ESPE, St. Paul, MN, USA) will be applied homogeneously to the surface with a disposable micro-brush. The cavity will be gently brushed with a faint air jet, allowing solvent evaporation, and light-cured for 10 s with an LED light (Smart Lite OS, Dentsply Indústria e Comércio Ltda., Rio de Janeiro/RJ - Brasil), with 1270 mW/cm2 of power density.

The class I teeth cavities will be restored with 2 mm increments of composite resin, by using a steel instrument (XTS Goldstein Flexi-Thin Mini #3, Hu-Friedy, Rio de Janeiro, RJ), and light-cured for 20 s, with the same light source and power density.

The finishing and polishing procedures will be performed after seven days, using fine diamond and multilaminated burs, followed by a one step polishing system Pogo (Dentsply, Caulk, USA). These procedures will be performed using a slow-speed hand piece with water spray. The disks, burs, and points will be discarded after each use.

For teeth assigned to the control group (NSS), they will be treated with finishing and polishing procedures only. Teeth included in SS group will be covered using a nanotechnology liquid polish system (Lasting Touch, Dentsply Caulk, Milford, DE, USA) applied as per the manufacturer's directions after finishing and polishing.. For this application, the composite surface and 1 mm external limit will be etched with a 37% acid phosphoric acid gel for 30 s and thoroughly rinse. The excess water will be removed with a mild oil free air stream, as per the manufacturer's instructions. Utilizing a disposable micro brush, a uniform layer of low-viscosity agent will be applied over the etched area, gently air brushed for 15 s and light-cured with the same light source.

The quality of the restorations will be rated according to the U.S. Public Health System/Ryge criteria. Two independent experienced examiners assessed the restorations. Restorations will bee calibrated according to Cohen's Kappa. Where disagreement occurred during evaluation, a consensus will be obtained among the examiners. It will be a double-blind evaluation, as neither examiner nor patients knew the treatment under evaluation. Examinations will be performed directly using mirror and probe. The evaluations will obtained at baseline (1 to 2 weeks after insertion) and 5 year after treatment. The parameters included will be marginal discoloration, anatomic form, secondary caries and marginal integrity. Data will be statistically analyzed using the McNemar's test (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Good oral hygiene;
* Having a class I caries lesion or unsatisfactory restoration in at least two posterior teeth (molar or premolar);
* Be in agreement and sign the consent form.

Exclusion Criteria:

* Patients with a proximal caries lesion;
* Presence of periodontal disease;
* Presence of symptomatic restored or non restored teeth indicating irreversible pulpal pathology;
* Presence of an abnormal occlusion or the absence of antagonist teeth;
* Presence of exposure of pulpal tissue;
* Presence of extended or large cavities.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Resin composite Longevity | baseline
  A clinical evaluation will be performed by two experienced operators using modified USPHS (United States Public Health service) at baseline, before the treatment. The parameters included will be marginal discoloration, anatomic form, secondary caries and marginal integrity.

SECONDARY OUTCOMES:
Resin composite longevity | 5-year
  A clinical evaluation will be performed by two experienced operators using modified USPHS (United States Public Health service) at 5 years after treatment. The parameters included will be marginal discoloration, anatomic form, secondary caries and marginal integrity.